CLINICAL TRIAL: NCT02215616
Title: A Multicenter, Multinational, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Laquinimod (0.5, 1.0 and 1.5 mg/Day) as Treatment in Patients With Huntington's Disease
Brief Title: A Clinical Study in Participants With Huntington's Disease (HD) to Assess Efficacy and Safety of Three Oral Doses of Laquinimod
Acronym: LEGATO-HD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TV5600-CNS-20007; 2014-000418-75 (EudraCT Number)
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — laquinimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive 3 capsules of matching laquinimod placebo, orally once daily for 52 weeks.
  Interventions: Drug: Placebo
- Laquinimod 0.5 mg (Experimental): Participants will receive 1 capsule of laquinimod 0.5 milligrams (mg) and 2 capsules of matching placebo, orally once daily for 52 weeks.
  Interventions: Drug: Laquinimod; Drug: Placebo
- Laquinimod 1.0 mg (Experimental): Participants will receive 2 capsule of laquinimod 0.5 mg (total 1.0 mg laquinimod) and 1 capsule of matching placebo, orally once daily for 52 weeks.
  Interventions: Drug: Laquinimod; Drug: Placebo
- Laquinimod 1.5 mg (Experimental): Participants will receive 3 capsules of laquinimod 0.5 mg (total 1.5 mg laquinimod), orally once daily.
  Note: The treatment of this high dose arm was discontinued as of 10 January 2016.
  Interventions: Drug: Laquinimod

INTERVENTIONS:
Drug: Laquinimod — Laquinimod capsules will be administered as per the dose and schedule specified in the respective arms.
  Arms: Laquinimod 0.5 mg; Laquinimod 1.0 mg; Laquinimod 1.5 mg
Drug: Placebo — Matching laquinimod placebo will be administered as per the schedule specified in the respective arms.
  Arms: Laquinimod 0.5 mg; Laquinimod 1.0 mg; Placebo

SUMMARY:
The primary objective of this study is to assess the efficacy of laquinimod as treatment in participants with HD after 52 weeks using the Unified Huntington's Disease Rating Scale Total Motor Score (UHDRS-TMS or TMS).

ELIGIBILITY:
Inclusion Criteria:

* Documentation of prior positive genetic testing for HD, or a clinical diagnosis of symptomatic HD.
* Presence of 36-49 cytosine-adenosine-guanine (CAG) repeats, inclusive, in the huntingtin gene based on centralized CAG testing during screening.
* Male or female between 21-55 years of age, inclusive, with an onset of HD at or after 18 years of age.
* Women of child-bearing potential (women who are not post menopausal or who have undergone surgical sterilization) must practice an acceptable method of birth control for 30 days before taking the study treatment, and 2 acceptable methods of birth control during all study duration and until 30 days after the last dose of treatment was administered.
* A sum of greater than (>) 5 points on the UHDRS-TMS at the screening visit.
* Able and willing to provide written informed consent prior to any study related procedure being performed at the screening visit. Participants with a legal guardian should be consented according to local requirements.
* Willing to provide a blood sample for genomic CAG analysis at the screening visit.
* Willing and able to take oral medication and able to comply with the study specific procedures.
* Ambulatory, being able to travel to the study center, and judged by the investigator as likely to be able to continue to travel for the duration of the study.
* Availability and willingness of a caregiver, informant, or family member to provide input at study visits assessing Clinician's Interview-Based Impression of Change (CIBIC)-Plus, Clinical Dementia Rating - Sum of Boxes (CDR-SB), Problem Behaviors Assessment-Short form (PBA-s) and Huntington's Disease Quality of Life (HD-QoL). A caregiver is recommended to be someone who attends to the participant at least 2 to 3 times per week for at least 3 hours per occasion, and the suitability of the caregiver should be judged by the investigator.
* For participants taking allowed antidepressant medication, the dosing of medication must have been kept constant for at least 30 days before baseline and must be kept constant during the study.

  * Additional criteria may apply, please contact the investigator for more information.

Exclusion Criteria:

* Use of immunosuppressive agents, or cytotoxic agents, including cyclophosphamide and azatioprine within 12 months prior to screening.
* Previous use of laquinimod.
* Use of moderate/strong inhibitors of cytochrome P450 (CYP)3A4 within 2 weeks prior to randomization.
* Use of inducers of CYP3A4 within 2 weeks prior to randomization.
* Pregnant or breastfeeding.
* Participants with a clinically significant or unstable medical or surgical condition that may put the participant at risk when participating in the study or may influence the results of the study or affect the participant's ability to take part in the study, as determined by medical history, physical examinations, electrocardiogram (ECG), or laboratory tests. Such conditions may include:

  * A major cardiovascular event (for example; myocardial infarction, acute coronary syndrome, de-compensated congestive heart failure, pulmonary embolism, coronary revascularization) that occurred prior to randomization.
  * Any acute pulmonary disorder.
  * A central nervous system (CNS) disorder other than HD that may jeopardize the participant's participation in the study, including such disorders that are demonstrated on the baseline MRI (based on local read).
  * A gastrointestinal disorder that may affect the absorption of study medication.
  * Acute or chronic renal disease including acute kidney injury (AKI).
  * Any form of acute or chronic liver disease.
  * Known human immunodeficiency virus (HIV) positive status. Participants will undergo an HIV test at screening per local requirements, if applicable.
  * Any malignancies, excluding basal cell carcinoma, in the 5 years prior to randomization.
* Any clinically significant, abnormal, screening laboratory result which in the opinion of the investigator, affects the participant' suitability for the study or puts the participant at risk if he/she enters the study.
* Unsuitable for MRI (for example; claustrophobia, metal implants).
* Alcohol and/or drug abuse within the 12 months prior to screening, as defined by Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition Text Revision (DSM IV TR) criteria for substance abuse.
* Participants with active suicidal ideation during the past month as measured by a most severe suicide ideation score of 4 (Active Suicidal Ideation with Some Intent to Act, without Specific Plan) or 5 (Active Suicidal Ideation with Specific Plan and Intent) on the baseline screening Columbia-Suicide Severity Rating Scale (C-SSRS) or participants who answer "Yes" on any of the 5 C-SSRS Suicidal Behavior Items (actual attempt, interrupted attempt, aborted attempt, preparatory acts, or behavior) if the attempt or acts were performed within 1 year of screening, or participants who, in the opinion of the investigator, present a serious risk of suicide.
* Participants with known intracranial neoplasms, vascular malformations, or intracranial hemorrhage.
* Known drug hypersensitivity that would preclude administration of laquinimod or placebo, such as hypersensitivity to mannitol, meglumine or sodium stearyl fumarate.
* Swallowing difficulties that would preclude administration of laquinimod or placebo capsules.
* Treatment with any investigational product within 30 days of screening or participants planning to participate in another clinical study assessing any investigational product during the study. Participants in non-interventional and/or observational studies will not be excluded from participating in this study.
* Treatment with tetrabenazine within 30 days of the study baseline visit.
* Treatment with antipsychotic medication within 30 days of the study baseline visit.

  * Additional criteria may apply, please contact the investigator for more information

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 352 (Actual)
Dates: Start 2014-10-28 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (16):
  - Teva Investigational Site 12566, La Jolla, California
  - Teva Investigational Site 12565, Los Angeles, California
  - Teva Investigational Site 12567, San Francisco, California
  - Teva Investigational Site 12575, Englewood, Colorado
  - Teva Investigational Site 13490, Tampa, Florida
  - Teva Investigational Site 13326, Iowa City, Iowa
  - Teva Investigational Site 12568, Wichita, Kansas
  - Teva Investigational Site 12574, Baltimore, Maryland
  - Teva Investigational Site 12571, Golden Valley, Minnesota
  - Teva Investigational Site 12572, St Louis, Missouri
  - Teva Investigational Site 12570, New York, New York
  - Teva Investigational Site 12569, Rochester, New York
  - Teva Investigational Site 13489, Memphis, Tennessee
  - Teva Investigational Site 13325, Nashville, Tennessee
  - Teva Investigational Site 12815, Houston, Texas
  - Teva Investigational Site 12576, Kirkland, Washington
- Canada (4):
  - Teva Investigational Site 11080, Vancouver, British Columbia
  - Teva Investigational Site 11118, Ottawa, Ontario
  - Teva Investigational Site 11079, Toronto, Ontario
  - Teva Investigational Site 11124, Edmonton
- Teva Investigational Site 54108, Prague, Czechia
- Germany (6):
  - Teva Investigational Site 32480, Berlin
  - Teva Investigational Site 32482, Bochum
  - Teva Investigational Site 32618, Erlangen
  - Teva Investigational Site 32483, München
  - Teva Investigational Site 32481, Münster
  - Teva Investigational Site 32479, Ulm
- Italy (5):
  - Teva Investigational Site 30168, Bologna
  - Teva Investigational Site 30098, Milan
  - Teva Investigational Site 30100, Milan
  - Teva Investigational Site 30097, Napoli
  - Teva Investigational Site 30099, San Giovanni Rotondo
- Teva Investigational Site 38066, Leiden, Netherlands
- Teva Investigational Site 36026, Lisbon, Portugal
- Russia (3):
  - Teva Investigational Site 50379, Kazan'
  - Teva Investigational Site 50380, Moscow
  - Teva Investigational Site 50381, Nyznij Novgorod
- Spain (6):
  - Teva Investigational Site 31185, Barakaldo
  - Teva Investigational Site 31097, Barcelona
  - Teva Investigational Site 31110, Barcelona
  - Teva Investigational Site 31186, Burgos
  - Teva Investigational Site 31131, Madrid
  - Teva Investigational Site 31187, Seville
- United Kingdom (10):
  - Teva Investigational Site 34176, Aberdeen
  - Teva Investigational Site 34177, Birmingham
  - Teva Investigational Site 34194, Liverpool
  - Teva Investigational Site 34179, London
  - Teva Investigational Site 34209, London
  - Teva Investigational Site 34204, London
  - Teva Investigational Site 34203, London
  - Teva Investigational Site 34175, Manchester
  - Teva Investigational Site 34215, Newcastle upon Tyne
  - Teva Investigational Site 34216, Sheffield

REFERENCES:
- [Derived] Reilmann R, Anderson KE, Feigin A, Tabrizi SJ, Leavitt BR, Stout JC, Piccini P, Schubert R, Loupe P, Wickenberg A, Borowsky B, Rynkowski G, Volkinshtein R, Li T, Savola JM, Hayden M, Gordon MF; LEGATO-HD Study Group. Safety and efficacy of laquinimod for Huntington's disease (LEGATO-HD): a multicentre, randomised, double-blind, placebo-controlled, phase 2 study. Lancet Neurol. 2024 Mar;23(3):243-255. doi: 10.1016/S1474-4422(23)00454-4. Epub 2024 Jan 24. PMID 38280392
- [Derived] Ehrnhoefer DE, Caron NS, Deng Y, Qiu X, Tsang M, Hayden MR. Laquinimod decreases Bax expression and reduces caspase-6 activation in neurons. Exp Neurol. 2016 Sep;283(Pt A):121-8. doi: 10.1016/j.expneurol.2016.06.008. Epub 2016 Jun 11. PMID 27296315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 468 participants were screened, of whom 116 participants were screen failures and 352 participants were enrolled. Of 352 enrolled participants, 123 participants were randomized in 1:1:1:1 ratio to receive laquinimod 0.5, 1.0, 1.5 milligrams/day (mg/day), or matching placebo prior to 10 January 2016.
Pre-assignment Details: As of 10 January 2016; following recommendation of Data Safety Monitoring Board (DSMB), treatment of laquinimod 1.5 mg dose arm was discontinued as a proactive safety measure. After 10 January 2016; additional eligible participants, who were enrolled, were randomized in 1:1:1 ratio to receive laquinimod 0.5 mg/day, 1.0 mg/day, or matching placebo.
Groups:
- Placebo: Participants received 3 capsules of matching laquinimod placebo, orally once daily for 52 weeks.
- Laquinimod 0.5 mg: Participants received 1 capsule of laquinimod 0.5 mg and 2 capsules of matching placebo, orally once daily for 52 weeks.
- Laquinimod 1.0 mg: Participants received 2 capsules of laquinimod 0.5 mg (total 1.0 mg laquinimod) and 1 capsule of matching placebo, orally once daily for 52 weeks.
- Laquinimod 1.5 mg: Participants received 3 capsules of laquinimod 0.5 mg (total 1.5 mg laquinimod), orally once daily. The treatment of this high dose arm was discontinued as of 10 January 2016.
Period: Overall Study
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1.0 mg | Laquinimod 1.5 mg
Started | 108 | 107 | 107 | 30
Received at Least 1 Dose of Study Drug | 108 | 107 | 106 | 29
Completed | 97 | 90 | 93 | 17
Not Completed | 11 | 17 | 14 | 13
Not completed — Sponsor requested to stop study drug | 0 | 0 | 1 | 4
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Adverse Event | 7 | 4 | 9 | 2
Not completed — Withdrawal by Subject | 1 | 8 | 2 | 5
Not completed — Non-compliance | 0 | 2 | 1 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 1
Not completed — Other than specified | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1.0 mg | Laquinimod 1.5 mg | Total
Number analyzed (Participants) | 108 | 107 | 107 | 30 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (7.76) | 43.3 (7.75) | 44.0 (7.83) | 45.5 (6.03) | 43.9 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 52 | 54 | 11 | 173
  Male | 52 | 55 | 53 | 19 | 179
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 104 | 103 | 105 | 28 | 340
  Black | 0 | 1 | 1 | 0 | 2
  Asian | 2 | 0 | 0 | 1 | 3
  Other | 0 | 1 | 0 | 0 | 1
  Missing | 2 | 2 | 1 | 1 | 6
Unified Huntington's Disease Rating Scale - Total Motor Score (UHDRS-TMS) [Mean (Standard Deviation); unit: units on a scale] — The UHDRS TMS assesses all the motor features of HD and includes maximal chorea, maximal dystonia, ocular pursuit, saccade initiation and velocity, dysarthria, tongue protrusion, finger tapping, hand pronation and supination, luria, rigidity, bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these was rated on a scale of 0 (normal motor function) to 4 (severely impaired motor function). TMS score is a sum of individual scores ranging from 0 (normal motor function) to 124 (severely impaired motor function). Lower TMS scores indicate better motor function. Population: 'Number analyzed' signifies participants evaluable for this parameter.
  units on a scale
    number analyzed (Participants) | 108 | 107 | 106 | 30 | 351
    (all) | 26.4 (14.63) | 24.0 (13.23) | 22.1 (10.74) | 26.8 (13.75) | 24.4 (13.12)
Normalized Caudate Volume [Mean (Standard Deviation); unit: milliliters (mL)] — Population: 'Number analyzed' signifies participants evaluable for this parameter.
  milliliters (mL)
    number analyzed (Participants) | 106 | 103 | 102 | 28 | 339
    (all) | 6.06 (1.857) | 5.78 (1.818) | 6.02 (1.781) | 5.39 (1.218) | 5.90 (1.781)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in UHDRS-TMS at Week 52
Description: UHDRS is a research tool developed by Huntington Disease (HD) Study Group to provide a uniform assessment of the clinical features and course of HD. Components of the full UHDRS assess motor function, cognition, behaviour, functional abilities, independence scale and total functional capacities. Motor function assessment includes TMS and Total Functional Capacity (TFC) score. The UHDRS TMS assesses all the motor features of HD and includes maximal chorea, maximal dystonia, ocular pursuit, saccade initiation and velocity, dysarthria, tongue protrusion, finger tapping, hand pronation and supination, luria, rigidity, bradykinesia, gait, tandem walking, and retropulsion pull test. Each of these was rated on a scale of 0 (normal motor function) to 4 (severely impaired motor function). TMS score is a sum of individual scores ranging from 0 (normal motor function) to 124 (severely impaired motor function). Lower TMS scores indicate better motor function.
Time Frame: Baseline, Week 52
Population: Full analysis set (FAS) included all participants in the ITT population (all randomized participants) who received at least 1 dose of study drug and had at least 1 post-baseline TMS assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1.0 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 98 | 92 | 95 | 4
units on a scale | 1.3 (8.00) | 1.4 (8.34) | 2.0 (7.27) | 11.0 (7.12)
Statistical Analysis 1: Comparison: Placebo vs Laquinimod 1.0 mg; Analysis was performed using Mixed Model Repeated Measures model (MMRM) with treatment group (3 levels: placebo, laquinimod 0.5 mg and laquinimod 1 mg), categorical week (4 levels: Weeks 4, 13, 26, and 52), treatment by week interaction, country, TMS baseline value and TMS baseline by week interaction as fixed effects. Unstructured variance-covariance structure was used in the initial model; Test type: Other; p = 0.4853, Mixed Models Analysis — Threshold for significance at 0.045 level; Least square (LS) mean difference = 0.78, 95% CI 2-sided [-1.42 to 2.98]

2. Secondary Outcome: Percent Change From Baseline in Caudate Volume (Brain Atrophy) at Week 52
Description: Brain atrophy was assessed using magnetic resonance imaging (MRI) measures of caudate volume. Caudate volume atrophy is a sensitive biomarker in very early HD and correlates with disease progression. Brain atrophy in the caudate refers to the shrinkage in volume, so that a decrease in volume is a positive value, while an increase in volume is a negative value. Percent change in caudate volume at Week 52 was calculated as the change in caudate volume since the baseline visit, divided by the baseline caudate volume and multiplied by 100.
Time Frame: Baseline, Week 52
Population: FAS included all participants in the ITT population (all randomized participants) who received at least 1 dose of study drug and had at least 1 post-baseline TMS assessment. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1.0 mg | Laquinimod 1.5 mg
Number analyzed (Participants) | 87 | 87 | 85 | 2
percent change | 5.13 (3.265) | 4.03 (3.275) | 3.14 (3.360) | 4.11 (0.598)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 56
Description: Safety analysis set included all participants who had received at least 1 dose of study drug.
Arm/Group | Placebo | Laquinimod 0.5 mg | Laquinimod 1.0 mg | Laquinimod 1.5 mg
All-Cause Mortality (participants affected / at risk) | 1/108 | 0/107 | 0/106 | 0/29
Serious Adverse Events (participants affected / at risk) | 8/108 | 7/107 | 5/106 | 1/29
Other Adverse Events (participants affected / at risk) | 62/108 | 69/107 | 58/106 | 19/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | Laquinimod 0.5 mg (N=107) | Laquinimod 1.0 mg (N=106) | Laquinimod 1.5 mg (N=29)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burn infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cluster headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=108) | Laquinimod 0.5 mg (N=107) | Laquinimod 1.0 mg (N=106) | Laquinimod 1.5 mg (N=29)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (10) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 12 (14) | 9 (11) | 3 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (10) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 7 (10) | 4 (7) | 2 (2)
Influenza (Infections and infestations) | 7 (9) | 8 (8) | 7 (7) | 0 (0)
Nasopharyngitis (Infections and infestations) | 19 (33) | 10 (12) | 10 (13) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 3 (5) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 6 (8) | 0 (0) | 1 (1) | 1 (3)
Fall (Injury, poisoning and procedural complications) | 9 (15) | 10 (12) | 5 (7) | 2 (6)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 2 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 4 (5) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 8 (10) | 6 (10) | 1 (1)
Blood folate decreased (Investigations) | 0 (0) | 1 (1) | 6 (6) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Pancreatic enzymes increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (7) | 4 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 7 (7) | 8 (12) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Chorea (Nervous system disorders) | 3 (4) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 7 (7) | 19 (22) | 14 (31) | 5 (5)
Anxiety (Psychiatric disorders) | 4 (4) | 3 (3) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 5 (7) | 0 (0) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 4 (4) | 2 (2) | 2 (2)
Irritability (Psychiatric disorders) | 4 (5) | 6 (7) | 3 (3) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4) | 6 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2016-02-16): https://cdn.clinicaltrials.gov/large-docs/16/NCT02215616/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT02215616/SAP_001.pdf